CLINICAL TRIAL: NCT04158869
Title: An Investigation of the Relationship Between Omega-3 Fatty Acid Nutrition and Mental Health in Children and Adolescents: A Case-control Study
Brief Title: An Investigation of the Relationship Between Omega-3 Fatty Acid Nutrition and Mental Health in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: n-3 case-control study
Record Dates: First submitted 2019-04-18; First posted 2019-11-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Major Depressive Disorder; Depression; Child Mental Disorder
Keywords: n-3 fatty acids; pediatric Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, hair, and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with pMDD, enrolled in the Investigator-initiated clinical trial IICT (ClinicalTrials.gov Identifier: NCT03167307)
- Controls: Controls matched to cases according to age, sex and school education

SUMMARY:
This is an observational case-control add-on study to an investigator-initiated clinical trial (IICT) (ClinicalTrials.gov Identifier: NCT03167307): Omega-3 fatty acids as firstline treatment in pediatric depression. A 36-week multi-centre, double-blind, placebo-controlled randomized superiority study.

This project will recruit a healthy control group matched for age and sex to a sub-group of patients with diagnosed pediatric major depressive disorder (pMDD) enrolled in the IICT. The aim is to investigate the relationship of n-3 FA intake and status with mental health in children and adolescents with and without diagnosed pMDD, and explore potential biochemical mechanisms underlying this relationship by measuring biomarkers related to n-3 FA metabolism, mental health and cognitive function.

DETAILED DESCRIPTION:
According to a recent school survey, one out of ten adolescents in Zurich have moderate to marked depressive symptoms. Early onset of paediatric major depressive disorder (pMDD) is a risk factor for chronic and recurrent forms of depression in adulthood (MDD). MDD is associated with difficulties in relationships, impaired school and work performance, and an increased risk of substance abuse. Furthermore, MDD is a major contributor to the burden of suicide and poor long-term health late in life. The emerging potential of n-3 polyunsaturated fatty acids (n-3 PUFAs), also known in short as omega-3 fatty acids (n-3 FAs), for the treatment of MDD is being investigated in several studies. Previous observational studies suggest a link between the consumption of n-3PUFA-rich food and the level of depressive symptoms. However, studies that investigated the potential beneficial effects of n-3 PUFA supplementation for the treatment of MDD compared with placebo showed inconsistent findings.

Primary objectives of this project are:

1. To determine the relationship of n-3 FA intake and status with mental health in children and adolescents with and without diagnosed pMDD.
2. To explore biochemical mechanisms underlying this relationship by measuring biomarkers related to n-3 FA metabolism, mental health, cognitive function, and potential pathways linking n-3 FA intake/status and brain health (e.g. immune system, gut microbiome-brain-axis).

Participants meeting the following criteria are eligible for the study:

Inclusion criteria:

* Participants of female and male sex
* Children aged 8 to ≤ 13 years or teenagers 13 to < 18 years at time of study entry
* Written informed assent of the subject and written informed consent from the subject's parents/legal representatives
* No present primary diagnosed psychiatric disorder according to the M.I.N.I. KID Test

Exclusion criteria:

* More than 4 weeks of regular n-3 FA supplementation
* Women who are self-reported pregnant or breast feeding
* Pre-existing neurological or medical conditions likely to be a risk factor for developing depressive symptoms

In a first step participants will be screened for in- and exclusion criteria. If participants can be included into the study we will

* Measure participant's mental health with behavioural and cognitive assessments
* Collect biological samples from participants (blood, urine, saliva, hair, and stool)

This study aims to recruit a total of 200 participants: 100 cases (from IICT) and 100 controls (recruited for this study).

There will be a total recruiting period of 18 months.

ELIGIBILITY:
For cases: participants enrolled in the IICT and therefore meeting the criterie for participation in the IICT will be selected.

For controls, participants fulfilling all of the following inlclusion criterie are eligible for the study

Inclusion Criteria:

* Participants of female and male sex
* Children aged 8 to ≤ 13 years or teenagers 13 to < 18 years at time of study entry
* Written informed assent of the subject (appendix informed consent forms) and written in formed consent form from the subjects' parents/legal representatives
* No present primary diagnosed psychiatric disorder according to the M.I.N.I. KID Test.
* No use of chronic medication
* Able to communicate in German; degree of understanding sufficient to comply with trial procedure

Exclusion Criteria:

* More than 4 weeks of regular n-3 FA supplementation (>2 daily capsules standard strength providing > 600 mg combined EPA/DHA) within the last 6 months.
* Women who are self-reported pregnant or breast feeding.
* Self-reported pre-existing neurological (such as e.g. brain tumour, temporal lobe epilepsy, HIV encephalopathy) or medical conditions (ICD-10 F06-F07) likely to be a risk factor for developing depressive symptoms
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children/adolescents in German speaking Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
n-3 fatty acid intake | 6 months
  Estimation of dietary omega-3 intake with a validated self-reported Omega-3 Food Questionnaire
n-3 fatty acid status | 1 day
  Measurement of relative amount of n-3 fatty acids
Pediatric depressive symptoms | 2 weeks
  Quantification of depressive symptoms with "Children's Depression Rating Scale - Revised" (CDRS-R) total score; Scale from 17 to >72; values >40 rated as moderate depression

SECONDARY OUTCOMES:
Fatty acid metabolism | 1 day
  Measurement of lipid mediators
Biomarkers related to brain health | 1 day
  Measurement of brain-derived neurotrophic factor (BDNF), kynurenine pathway metabolites, and monoamine neurotransmitters
Biomarkers related to systemic inflammation | 1 day
  Measurement of C-reactive Protein (CRP), alpha-1-acid glycoprotein, and cytokines
Biomarkers related to gut microbiota | 1 day
  Measurement of
  * gut microbiome composition with 16S rRNA sequencing
  * Faecal calprotectin
  * Intestinal fatty acid binding protein
Biomarkers related to nutritional status | 1 day
  Measurement of iron and iodine status

OTHER OUTCOMES:
Verbal learning and memory test (VLMT) | 1 day
  Differences in scores between cases and controls
Behavior Rating Inventory of Executive Function (BRIEF) | 1 day
  Differences in the overall score between cases and controls
Digit span measured by the Wechsler Intelligence Scale for children (WISC-IV) | 1 day
  Differences in scores between cases and controls
Emotion recognition measured with the Amsterdam Neuropsychological Task (ANT) program | 1 day
  Differences in scores between cases and controls
Attentional flexibility measured with the shifting attentional set of the Amsterdam Neuropsychological Task (ANT) program | 1 day
  Differences in reaction times between cases and controls
Regensburg Word Fluency Test (RWT) | 1 day
  Differences in scores between cases and controls
Reynolds Intellectual Assessment Scales (RIAS) | 1 day
  Differences in scores between cases and controls
Suicidal ideation Questionnaire (SIQ) | 1 month
  Differences in scores between cases and controls
Scale of Impulsivity and Emotion Dysregulation (IES-27) | 1 month
  Differences in scores between cases and controls
Childhood Trauma Questionnaire (CTQ) | 1 day
  Differences in scores between cases and controls
Strenght and Difficulty Questionnaire (SDQ) | 1 day
  Differences in scores between cases and controls
Perceived Stress Scale (PSS-10) | 1 month
  Differences in scores between cases and controls
Children's Depression Inventory (DIKJ) | 1 month
  Differences in scores between cases and controls
Connor Davidson Resilience Scale (CDRS) | 1 month
  Differences in scores between cases and controls
Beck Anxiety Inventory (BAI) | 1 month
  Differences in scores between cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Berger, Dr. med., Study Chair — Psychiatrische Universitätsklinik Zürich; Jeannine Baumgartner, Dr., Principal Investigator — Swiss Federal Institute of Technology; Isabelle Herter-Aeberli, Dr., Principal Investigator — Swiss Federal Institute of Technology; Michael B Zimmermann, Dr. med., Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- ETH Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
A BioBank will be established. Access to the Biobank can be requested upon completion of the IICT and the add-on study contacting the principal investigator Dr. Jeannine Baumgartner
Supporting Information: Study Protocol, SAP
Time Frame: upon study completion of the IICT and the add-on study.